CLINICAL TRIAL: NCT06511999
Title: Feasibility and Validation of Continuous Measurement of Jugular Venous Oxygen Saturation in Comatose Patients After Cardiac Arrest
Brief Title: Continuous Jugular Venous Oxygen Saturation (SjO2) Measurement After Cardiac Arrest
Status: Recruiting | Type: Observational
Sponsor: Byron Drumheller (Other)
Responsible Party: Sponsor-Investigator, Byron Drumheller, Assistant Professor of Emergency Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Other Study IDs: STUDY24040111
Record Dates: First submitted 2024-07-15; First posted 2024-07-22 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-07

CONDITIONS: Cardiac Arrest
Keywords: Jugular venous oxygen saturation; Neuromonitoring
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be withdrawn from the jugular venous catheter at 0, 24, 48 and 72 hours after insertion for measurement of protein biomarkers associated with secondary brain injury after cardiac arrest.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Comatose participants resuscitated from cardiac arrest: Participants successfully resuscitated from cardiac arrest that are comatose (motor glasgow coma scale <= 4) upon initial assessment will undergo jugular venous oxygen saturation (SjO2) monitoring with the study device [PediaSat Oximetry Catheter, Edwards Lifesciences Corp, Irvine, CA].
  Interventions: Device: Continuous SjO2 monitoring with a PediaSat Oximetry Catheter; Diagnostic Test: Intermittent SjO2 monitoring with a PediaSat Oximetry Catheter

INTERVENTIONS:
Device: Continuous SjO2 monitoring with a PediaSat Oximetry Catheter — The PediaSat Oximetry Catheter is capable of continuous, indwelling measurement of venous oxygen saturation, which is displayed on a bedside monitor connected by an optical cable. Enrolled participants will undergo continuous SjO2 measurement for 72 hours. Clinical care will not be directed by the continuous SjO2 values.
Diagnostic Test: Intermittent SjO2 monitoring with a PediaSat Oximetry Catheter — The PediaSat Oximetry Catheter is also capable of intermittent blood sampling enabling measurement of SjO2 on a laboratory blood gas analyzer. Enrolled participants will undergo intermittent SjO2 measurement every 4-6 hours for 72 hours. Clinical care will be directly by the intermittent values.

SUMMARY:
Patients successfully resuscitated from sudden cardiac arrest are often comatose, having suffered a period of low blood flow and oxygen delivery to the brain. They are also at risk of suffering further brain injury during the immediate period after resuscitation, in which the brain's normal regulatory functions are impaired. To diagnose and treat secondary brain injury in comatose patients after cardiac arrest, doctors use a variety of neurological monitoring techniques. One of these methods involves measuring the oxygen saturation of blood going into and out of the brain to determine whether the brain is receiving and utilizing oxygen in an optimal manner. The oxygen saturation of blood exiting the brain is called the jugular venous oxygen saturation (SjO2). It is measured by inserting a catheter into the jugular vein in the neck and sampling blood as it exits the skull. The blood sample is sent to the hospital laboratory and the oxygen saturation is measured on a blood gas machine. This method of SjO2 measurement has limitations, particularly that blood must be taken out of the patient and sent to the lab for analysis, which can only be done feasibly every few hours. Special catheters exist that can measure the oxygen saturation of blood passing by the tip of the catheter inside the patient on a second-by-second basis, without needing to withdraw blood and send it to the laboratory. With such rapidly available data, doctors may be able to better diagnose and treat brain oxygen abnormalities in post cardiac arrest patients.

In this study, the investigators plan to determine the accuracy of an existing, Food and Drug Administration (FDA)-cleared catheter capable of continuous, indwelling measurement of venous blood oxygen saturation for SjO2 monitoring in comatose patients early after cardiac arrest. The SjO2 measurements from the study catheter will be compared with standard SjO2 measurements made by withdrawing blood and analyzing it in the laboratory to determine if the new catheter is accurate. The investigators will also collect blood samples using the study catheter to measure levels of specific proteins that indicate damage to brain tissue. The study will enroll 25 participants admitted to the intensive care unit at one hospital cared for by a group of doctors that specialize in the neurological care of patients after cardiac arrest. The investigators hypothesize that the study catheter will accurately measure SjO2 compared to the standard laboratory method.

DETAILED DESCRIPTION:
Patients who achieve return of spontaneous circulation (ROSC) after sudden cardiac arrest and remain comatose are at high risk of secondary brain injury that may prevent or worsen the quality of neurological recovery. Current treatments that attempt to mitigate the extent of secondary brain injury include targeted temperature management (TTM), maintenance of adequate blood pressure and gas exchange (oxygen and carbon dioxide), and antiepileptic treatment of seizures and other hyperexcitable patterns detected on electroencephalographic (EEG) monitoring. Multiple recent large-scale clinical trials comparing different magnitudes of such therapies (mild hypothermia vs. controlled normothermia or fever prevention, aggressive antiseizure treatment of rhythmic/periodic patterns vs. no treatment) or resuscitation targets (oxygen, carbon dioxide, and blood pressure goals) did not detect improvement in neurologic outcome with the hypothesized superior interventions. Research from the investigators and others suggests that between-patient heterogeneity in patterns and severity of hypoxic-ischemic brain injury (HIBI) after cardiac arrest may explain the repeated failure to find a population-level benefit of any particular one-size-fits-all therapy: individual patients exhibit differing pathophysiology and may respond best to different neuroprotective interventions.

To tailor potential neuroprotective treatments to individual patients, doctors must be able to detect and characterize neurological pathophysiology and treatment responsiveness in real time. This requires use of one or more prospective neuromonitoring modalities, including measurement of jugular venous oxygen saturation (SjO2). Measurement of SjO2 involves inserting a catheter retrograde into the internal jugular vein and determining the oxygen saturation of blood just after it leaves the skull. By comparing the SjO2 with the saturation of arterial blood (SaO2) entering the brain, measured from a large artery, the percentage of oxygen extracted by the brain can be determined (SaO2 - SjO2). This is akin to measuring central venous oxygen saturation (ScvO2) in various types of circulatory shock. Measurement of SjO2 early after cardiac arrest provides information on the balance between brain-specific oxygen supply, utilization, and demand. Identification of abnormal brain oxygen balance during this time period in which secondary brain injury is most likely to occur can trigger and guide potentially corrective therapies.

The Post Cardiac Arrest Service (PCAS) at UPMC Presbyterian uses SjO2 monitoring in comatose patients after cardiac arrest as part of routine prognostic and therapeutic purposes for the first 72 hours of hospitalization. Prior research has shown a significant association between elevated mean SjO2 (>75%) during the early post-arrest period and poor outcomes. It is hypothesized that this represents either poor brain oxygen extraction resulting from abnormalities in diffusion through peri-neuronal tissue or impaired mitochondrial oxygen uptake and utilization, leading to elevated oxygen saturation/content in venous blood leaving the injured brain. Preliminary case series by the investigators and Hoiland et al. have shown that some patients with elevated SjO2 exhibit a decrease in SjO2, and concomitant increase in brain oxygen utilization, after treatment with hypertonic saline (HTS), suggesting that abnormal oxygen diffusion due to perivascular edema plays some part in the pathophysiology of post-arrest HIBI.

The ability to detect and act upon abnormal brain oxygen balance, particularly oxygenation changes that may result from potential neuroprotective interventions, is limited by current SjO2 measurement technology. Presently, SjO2 is measured by withdrawing blood from a single lumen, 3-4 French, 10-15 cm-long catheter on an intermittent basis every 4-6 hours and calculating venous oxygen saturation from the blood sample on a blood gas analyzer in the hospital laboratory. As a result, SjO2 data granularity is limited by the practical frequency of blood draws and lab result turn-around time. However, vascular catheter technology allowing for continuous, in-dwelling measurement of venous blood oxygen saturation via spectrophotometry exists and is routinely used to monitor central venous oxygen saturation (ScvO2) and mixed venous oxygen saturation (SvO2) in patients with cardiogenic shock. Specifically, an FDA-cleared, continuous venous oximetry-enabled, central venous catheter [PediaSat™ Oximetry Catheter, Edwards Lifesciences Corp, Irvine, CA] [triple lumen, 5.5 French, 15 cm] is currently used for measurement of ScVO2 in pediatric patients with cardiogenic or septic shock. This catheter also allows for intermittent blood sampling. The investigators seek to translate this existing continuous venous oximetry technology for use in the measurement of SjO2. To do so, the investigators plan to perform a prospective, observational, case series study to determine the feasibility and accuracy of continuous measurement of SjO2 with the PediaSat™ Oximetry Catheter , compared to the standard technique of measurement via blood sampling analysis on a laboratory blood gas machine, in comatose participants at risk of secondary brain injury after cardiac arrest. The investigators also plan to demonstrate the feasibility of obtaining and storing jugular blood samples using the continuous SjO2 catheter for future biomarker analysis.

ELIGIBILITY:
Inclusion Criteria:

• Adults (>=18 years old) resuscitated from out-of-hospital or in-hospital cardiac arrest who remain comatose (motor Glasgow coma scale <=4) for at least 30 minutes when examined off sedation/neuromuscular blockade.

Exclusion Criteria:

* Cardiac arrest due to traumatic brain injury, intracranial bleeding, or ischemic stroke
* Cervical spine fracture
* Need for immediate prone positioning for severe hypoxemic respiratory failure
* Marked hemodynamic instability precluding priority of any neuromonitoring (multiple recurrent cardiac arrests, norepinephrine equivalents > 1.5 mcg/kg/min)
* Moribund neurological status based upon initial clinical, radiographic and historical assessment (e.g. diffuse cerebral edema or herniation on head computed tomography)
* Pregnancy
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients successfully resuscitated from cardiac arrest
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-09-20 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Bias and percent error of continuous SjO2 measurements compared to intermittent SjO2 measurements, both obtained with the PediaSat Oximetry Catheter | From hospital presentation to 72 hours after admission
  The accuracy of SjO2 measurement with the PediaSat Oximetry Catheter will be determined by comparing the SjO2 measurements obtained from the study catheter with the gold standard of SjO2 measured on jugular venous blood simultaneously withdrawn from the catheter and analyzed on a blood gas machine. Each participant will have ~10-15 paired SjO2 measurements. The Bland-Altman method for assessing agreement between two methods of clinical measurement with multiple observations per participant will be utilized to calculate the bias between the mean differences of the continuous and intermittent techniques and the percent error of the continuous technique. Based on established accuracy requirements for similar continuous in-vivo measurements in critical care, a bias of <= ± 5 and a percent error of <= 30 will be considered successful.

SECONDARY OUTCOMES:
Proportion of participants in which the PediaSat Oximetry Catheter is successfully inserted and all intermittent and continuous SjO2 measurements are obtained | From hospital presentation to 72 hours after admission
  Feasibility will be measured by calculating the proportion of participants in which the PediaSat Oximetry Catheter is successfully inserted and SjO2 data is successfully collected for 72 hours, as determined by routine clinical care. For an individual participant to achieve feasibility, the catheter must be correctly inserted and all intermittent and continuous SjO2 measurements ordered as part of clinical care must be measured successfully. The study goal is for >= 75 percent of participants to achieve feasibility.
Proportion of participants in which all study blood samples are collected, processed, and stored successfully. | From hospital presentation to 72 hours after admission
  Feasibility of obtaining serial jugular venous blood samples during the first 72 hours of post-arrest care and storage of plasma for subsequent biomarker analysis will be measured by calculating the proportion of participants in which all 4 study blood samples are collected, processed, and successfully stored. The study goal is for >= 75 percent of participants to achieve feasibility.

CONTACTS AND LOCATIONS:
Overall Officials: Byron Drumheller, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Skrifvars MB, Sekhon M, Aneman EA. Monitoring and modifying brain oxygenation in patients at risk of hypoxic ischaemic brain injury after cardiac arrest. Crit Care. 2021 Aug 31;25(1):312. doi: 10.1186/s13054-021-03678-3. PMID 34461973
- [Background] Le Roux P, Menon DK, Citerio G, Vespa P, Bader MK, Brophy G, Diringer MN, Stocchetti N, Videtta W, Armonda R, Badjatia N, Bosel J, Chesnut R, Chou S, Claassen J, Czosnyka M, De Georgia M, Figaji A, Fugate J, Helbok R, Horowitz D, Hutchinson P, Kumar M, McNett M, Miller C, Naidech A, Oddo M, Olson D, O'Phelan K, Provencio JJ, Puppo C, Riker R, Roberson C, Schmidt M, Taccone F. The International Multidisciplinary Consensus Conference on Multimodality Monitoring in Neurocritical Care: a list of recommendations and additional conclusions: a statement for healthcare professionals from the Neurocritical Care Society and the European Society of Intensive Care Medicine. Neurocrit Care. 2014 Dec;21 Suppl 2(Suppl 2):S282-96. doi: 10.1007/s12028-014-0077-6. PMID 25501689
- [Background] Hoiland RL, Ainslie PN, Wellington CL, Cooper J, Stukas S, Thiara S, Foster D, Fergusson NA, Conway EM, Menon DK, Gooderham P, Hirsch-Reinshagen V, Griesdale DE, Sekhon MS. Brain Hypoxia Is Associated With Neuroglial Injury in Humans Post-Cardiac Arrest. Circ Res. 2021 Aug 20;129(5):583-597. doi: 10.1161/CIRCRESAHA.121.319157. Epub 2021 Jul 21. PMID 34287000
- [Background] Sekhon MS, Ainslie PN, Menon DK, Thiara SS, Cardim D, Gupta AK, Hoiland RL, Gooderham P, Griesdale DE. Brain Hypoxia Secondary to Diffusion Limitation in Hypoxic Ischemic Brain Injury Postcardiac Arrest. Crit Care Med. 2020 Mar;48(3):378-384. doi: 10.1097/CCM.0000000000004138. PMID 31789834
- [Background] Richter J, Sklienka P, Chatterjee N, Maca J, Zahorec R, Burda M. Elevated jugular venous oxygen saturation after cardiac arrest. Resuscitation. 2021 Dec;169:214-219. doi: 10.1016/j.resuscitation.2021.10.011. Epub 2021 Oct 19. PMID 34678332
- [Background] Bland JM, Altman DG. Statistical methods for assessing agreement between two methods of clinical measurement. Lancet. 1986 Feb 8;1(8476):307-10. PMID 2868172
- [Background] Howard L, Gopinath SP, Uzura M, Valadka A, Robertson CS. Evaluation of a new fiberoptic catheter for monitoring jugular venous oxygen saturation. Neurosurgery. 1999 Jun;44(6):1280-5. PMID 10371628
- [Background] Bland JM, Altman DG. Agreement between methods of measurement with multiple observations per individual. J Biopharm Stat. 2007;17(4):571-82. doi: 10.1080/10543400701329422. PMID 17613642